CLINICAL TRIAL: NCT05121285
Title: Distribution of FMT After Delivery by · Lower GI Endoscopy vs· Enema With and Without Positioning of the Patient
Brief Title: Distribution of FMT After Delivery by · Lower GI Endoscopy vs Enema With and Without Positioning of the Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 267433
Record Dates: First submitted 2021-11-03; First posted 2021-11-16 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2021-10

CONDITIONS: Fecal Microbiota Transplantation
MeSH Terms: interventions — Patient Positioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contrast fluid by lower GI endoscopy and enema with and without positioning (Experimental): There is a washout period of at least four weeks between the two interventions (delivery by lower GI endoscopy and enema)
  Interventions: Other: Delivery of contrast fluid by lower GI endoscopy; Other: Delivery of contrast fluid by enema with and without positioning

INTERVENTIONS:
Other: Delivery of contrast fluid by lower GI endoscopy — Each participant will receive one delivery of 440 ml contrast fluid by lower GI endoscopy to the cecum of the colon. The participants perform a bowel lavage using Sodiumpicosulphate/Magnesiumcitrate (Picoprep, Ferring) 24 hours before the delivery of contrast fluid. An colon X-ray is obtained within 10 minutes after the contrast fluid is delivered. The participants is in a supine position fram delivery and until the colon x-ray is obtained.
Other: Delivery of contrast fluid by enema with and without positioning — Each participant will receive one delivery of 440 ml contrast fluid by enema. The participants perform a bowel lavage using Sodiumpicosulphate/Magnesiumcitrate (Picoprep, Ferring) 24 hours before the delivery of contrast fluid. The enema procedure includes:
  1. The participant lies on his/her left side in neutral position when the enema is delivered
  2. X-ray of the colon is obtained with the participant lying on his/her back.
  3. The participant is positioned back to his/her left sided position and tilted in a Trendelenburg position. The position is held for two minutes
  4. The participant is turned to an abdominal position while the bed remains tilted in Trendelenburg position.
  5. Participant turne to the right side. When positioned the bed is tilted the opposite way (anti-Trendelenburg.) The position is held for two minutes.
  6. A second colon X-ray is obtained after the participants has rested for ten minutes in a supine neutral position

SUMMARY:
While delivery of an FMT-treatment to the cecum is visualized in a lower GI-endoscopy, it is uncertain whether delivery by enema distributes the FMT to the proximal segments of the colon. Positioning of the patient during the enema procedure may improve distribution to the proximal colon. Differences in distribution may explain the wide effect range and inferiority when enema is compared to delivery by lower GI endoscopy. Thus, in this study we will compare the distribution of FMT from delivery by lower GI endoscopy versus enema with and without positioning of the patient. We will use contrast fluid as a surrogate liquid for FMT to project the distribution on colon X-ray pictures. To our knowledge this is not done in any previous study.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for colonoscopy at the medical department at UNN Harstad
* Able to complete the positioning procedure during the enema

Exclusion Criteria:

* Confirmed malignancy
* Inflammatory bowel disease
* Referral highly suspicious of cancer, inflammatory bowel disease or obstructive GI disease
* Contraindications for rectal catheter insertion (including known damage to pelvic floor, sphincter or the pudendal nerve)
* Use of anticoagulants. Use of acetylsalicylic acid is allowed
* Symptomatic cardiovascular or lung disease
* Kidney failure
* Known allergic reaction to any component in Liquid Polibar Plus
* Pregnant, lactating or planning pregnancy
* Asthma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Proportion of cecum projection after CF delivery by lower GI endoscopy versus enema with positioning versus enema without positioning of the participants. | 10 minutes after contrast fluid delivery
  Two radiologist determine the projection each colon X-ray picture by identifying segments where the gut mucosa is coated with contrast fluid and/or segments with contrast fluid in the lumen. The radiologist is blinded to which delivery method is used.

SECONDARY OUTCOMES:
Proportion of transverse colon projection after CF delivery by the lower GI endoscopy versus enema with positioning versus enema without positioning of the participants. | 10-20 minutes after contrast fluid delivery
  Two radiologist determine the projection each colon X-ray picture by identifying segments where the gut mucosa is coated with contrast fluid and/or segments with contrast fluid in the lumen. The radiologist is blinded to which delivery method is used.

CONTACTS AND LOCATIONS:
Overall Officials: Peter H Johnsen, MD PhD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Harstad, Harstad, Troms, Norway

IPD SHARING:
Plan to Share IPD: Yes
Study protocol with statistical analysis plan will be uploaded to the ClinicalTrials.gov web site.
Supporting Information: Study Protocol, SAP
Time Frame: Within 2021

REFERENCES:
- [Derived] Skjevling LK, Hanssen HM, Valle PC, Goll R, Juul FE, Arlov O, Johnsen PH. Colonic distribution of FMT by different enema procedures compared to colonoscopy - proof of concept study using contrast fluid. BMC Gastroenterol. 2023 Oct 23;23(1):363. doi: 10.1186/s12876-023-02979-x. PMID 37872499